CLINICAL TRIAL: NCT07336004
Title: Breastfeeding: Influencing Determinants, Knowledge and Self-efficacy Among Lactating Mothers in Sohag Governorate
Brief Title: Breastfeeding: Influencing Determinants, Knowledge and Self-efficacy
Acronym: feeding
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Rahma Ibrahim Mahmoud, Assistant lecturer, Sohag University
Other Study IDs: Soh-Med--25-12-3MD
Record Dates: First submitted 2025-12-13; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Breastfeeding, Exclusive; Breastfeeding Initiation
Keywords: breastfeeding; Beastfeeding exclusivness
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- lactating mothers

SUMMARY:
Our study will assess the prevalence of exclusive breastfeeding and the determinants and assess knowledge and self efficacy of lactating mothers towards breastfeeding

ELIGIBILITY:
Inclusion criteria:

• The study will include lactating mothers with children from day zero to 24 months.

Exclusion criteria:

* Mothers with absolute contraindications to breastfeeding as the infant having classic galactosemia
* The mother having human immunodeficiency virus (HIV) will be excluded from the study.

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — the study concerned about lactating mothers
Study Population: lactating mothers
Sampling Method: Probability Sample
Enrollment: 380 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
timely initiation of breastfeeding | two years
  (expressed as the proportion of infants who first suckled within 1 hour after birth)
exclusive breastfeeding | two years
  expresses as the proportion of infants below 6 months who fed only on breast milk in the 24-hours preceding the survey to the total number of children in the same age group (< 6 months of age).

SECONDARY OUTCOMES:
Breastfeeding knowledge | two years
  Afan Oromo (AO) versions of the Breastfeeding Knowledge Questionnaire (BFKQ): The BFKQ-AO consists of 34 items asking about various optimal breastfeeding practices, with responses coded as correct or incorrect. It contained nine domains: advantage to baby, advantage to mothers, colostrum, breast milk expression, duration of feeding, problems with breastfeeding, breast engorgement, practical aspects of breastfeeding (Tengku Ismail and Sulaiman, 2010; Abdulahi et al., 2021)
Breastfeeding self-efficacy | two years
  The BSES-SF is a 14-item self-administered instrument (Amini et al., 2019) derived from the original 33-item BSES that measures breastfeeding confidence (Dennis, 2003). All items are preceded by the phrase ''I can always'' and rated on a 5-point Likert scale, ranging from 1 (not at all confident) to 5 (always confident). Total scores range from 14 to 70, with higher scores reflecting more significant levels of breastfeeding self-efficacy. The higher the score, the higher the level of breastfeeding self-efficacy.